CLINICAL TRIAL: NCT01692275
Title: Assessment of Chiropractic Treatment for Low Back Pain and Smoking Cessation in Military Active Duty Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Palmer College of Chiropractic (Other); Samueli Institute for Information Biology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2010-0782
Record Dates: First submitted 2012-09-06; First posted 2012-09-25 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Ice

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical Care + Chiropractic Care (Active Comparator): Medical care plus chiropractic manipulative therapy
  Interventions: Other: Medical Care + Chiropractic Care
- Conventional Medical Care Only (Active Comparator): Conventional medical care only
  Interventions: Other: Conventional Medical Care Only

INTERVENTIONS:
Other: Medical Care + Chiropractic Care — Patients will receive chiropractic spinal manipulative therapy plus conventional medical care. Medical may include the following: education about self-management, including maintaining activity levels as tolerated and local ice/heat application; pharmacologic management with the use of analgesics and anti-inflammatory agents; and additional therapies that may be applied for volunteers not responding to the initial interventions, including physical therapy and referral to a pain clinic.
  Other Names: spinal manipulative therapy; education self management medication heat and ice
  Arms: Medical Care + Chiropractic Care
Other: Conventional Medical Care Only — Conventional medical care may include the following: a focused history and physical examination; limited diagnostic imaging restricted to select volunteers (i.e., for example, those with radiculopathy); education about self-management, including maintaining activity levels as tolerated and local ice/heat application; pharmacologic management with the use of analgesics and anti-inflammatory agents; and additional therapies that may be applied for volunteers not responding to the initial interventions, including physical therapy and referral to a pain clinic.
  Arms: Conventional Medical Care Only

SUMMARY:
The purpose of this study is to evaluate the effectiveness of chiropractic manipulative therapy for pain management and improved function in active duty service members with low back pain that do not require surgery. The study will also measure the impact of a tobacco cessation program delivered to participants allocated to the chiropractic arm.

DETAILED DESCRIPTION:
Low back pain (LBP) is the most common cause of disability worldwide, but it is even more prevalent in active duty military personnel; more than 50% of all diagnoses resulting in disability discharges from the military across all branches are due to musculoskeletal conditions. LBP has been characterized as "The Silent Military Threat" because of its negative impact on mission readiness and the degree to which it compromises a fit fighting force. For these reasons, military personnel with LBP need a practical and effective treatment that relieves their pain and allows them to return to duty quickly, but also one that preserves function and military readiness, addresses the underlying causes of the episode and protects against re-injury. Currently a clear "gold standard" medical treatment for low back pain does not exist and studies show that evidence-based guidelines are rarely used in general practice. Thus, there is a need to consider innovative treatment options for chronic diseases such as LBP. Therefore the primary purpose of this study is to assess the effectiveness of chiropractic manipulative therapy (CMT) for pain management and improved function in active duty service members with orthopedic injuries or disorders of the low back that do not require surgery. This multi-site Phase II Clinical Comparative Effectiveness Trial is designed to rigorously compare the outcomes of CMT and conventional medical care (CMC) to CMC alone. Chiropractic treatment will include CMT plus ancillary physiotherapeutic interventions. CMC will be delivered following current standards of medical practice at each site. At each of the four participating sites, active military personnel, ages 18-50, who present with acute, sub-acute or chronic low back pain that does not require surgery will be randomized to one of the two treatment groups. Outcome measures include the Numerical Rating Scale for pain, the Roland-Morris Low Back Pain and Disability questionnaire, the Back Pain Functional Scale for assessing function, and the Global Improvement questionnaire for patient perception regarding improvement in function. Patient Expectation and Patient Satisfaction questionnaires will be used to examine volunteer expectations toward care and perceptions of that care. Pharmaceutical use and duty status data will also be collected. The PROMIS-29 will be utilized to compare the general health component and quality of life of the sample at baseline. In addition, doctors of chiropractic are well positioned to provide information to support tobacco cessation. Thus this clinical trial will include a nested study designed to measure the impact of a tobacco cessation program delivered by a doctor of chiropractic. The results from this randomized clinical trial, with a nested tobacco cessation intervention, will provide critical information regarding the health and mission-support benefits of chiropractic health care delivery for active duty service members in the military

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 (Inclusive)
* Diagnosis of acute, subacute or chronic low back pain
* Ability to provide voluntary written informed consent
* Active duty at one of the three participating military sites

Exclusion Criteria:

* LBP from other than somatic tissues as determined by history, examination and course (i.e., pain referred from visceral conditions)
* Co-morbid pathology or poor health conditions that may directly impact spinal pain
* Volunteers who have case histories and physical examination findings indicating other than average good health
* Bone and joint pathology contraindicating CMT (Chiropractic Manipulative Therapy)
* Volunteers with recent spinal fracture (within the last 8 weeks), recent spinal surgery (within the last 12 weeks), concurrent spinal or paraspinal tumor(s), spinal or paraspinal infection(s), inflammatory arthropathies and significant/severe osteoporosis will be referred for appropriate care
* Other contraindications for CMT of the lumbar spine and pelvis (i.e., unstable spinal segments, cauda equine syndrome)
* Pregnant or planning to become pregnant within 3 months
* Altered mental capacity as determined by the clinician
* Unable to speak English
* Use of manipulative care for any reason within the past month
* Unwilling to provide phone and electronic contact information
* Unable to confirm that they will not be transferred during the active phase of the study, i.e., deployment, receive orders for a distant duty assignment or training site or otherwise be absent from the current military site over the next 8 weeks (active study participation period).
* Does not agree to be enrolled regardless of group assignment
* PTSD Classification

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 750 (Actual)
Dates: Start 2012-09; Primary Completion 2016-11-28 (Actual); Study Completion 2016-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian D. Coulter, Ph.D., Principal Investigator — RAND
Locations (3):
- United States (3):
  - Naval Medical Center San Diego, San Diego, California
  - Naval Hospital Pensacola, Pensacola, Florida
  - Walter Reed National Military Medical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goertz CM, Long CR, Vining RD, Pohlman KA, Kane B, Corber L, Walter J, Coulter I. Assessment of chiropractic treatment for active duty, U.S. military personnel with low back pain: study protocol for a randomized controlled trial. Trials. 2016 Feb 9;17:70. doi: 10.1186/s13063-016-1193-8. PMID 26857706
- [Background] Goertz CM, Long CR, Vining RD, Pohlman KA, Walter J, Coulter I. Effect of Usual Medical Care Plus Chiropractic Care vs Usual Medical Care Alone on Pain and Disability Among US Service Members With Low Back Pain: A Comparative Effectiveness Clinical Trial. JAMA Netw Open. 2018 May 18;1(1):e180105. doi: 10.1001/jamanetworkopen.2018.0105. PMID 30646047
- [Derived] Shannon ZK, Long CR, Chrischilles E, Goertz C, Wallace R, Casteel C, Carnahan RM. Secondary causal mediation analysis of a pragmatic clinical trial to evaluate the effect of chiropractic care for US active-duty military on biopsychosocial outcomes occurring through effects on low back pain interference and intensity. BMJ Open. 2024 Nov 19;14(11):e083509. doi: 10.1136/bmjopen-2023-083509. PMID 39566948

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medical Care + Chiropractic Care | Conventional Medical Care Only
Started | 375 | 375
Completed | 309 | 316
Not Completed | 66 | 59
Not completed — Lost to Follow-up | 57 | 48
Not completed — Withdrawal by Subject | 9 | 11

BASELINE CHARACTERISTICS:
Groups:
- Site: WRNMMC - UMC: Site: Walter Reed National Military Medical Center (WRNMMC) Conventional medical care only/Usual Medical Care (UMC)
  Conventional Medical Care Only: Conventional medical care may include the following: a focused history and physical examination; limited diagnostic imaging restricted to select volunteers (i.e., for example, those with radiculopathy); education about self-management, including maintaining activity levels as tolerated and local ice/heat application; pharmacologic management with the use of analgesics and anti-inflammatory agents; and additional therapies that may be applied for volunteers not responding to the initial interventions, including physical therapy and referral to a pain clinic.
- Site: WRNMMC - UMC + Chiropractic Care: Site: Walter Reed National Military Medical Center (WR)
  Medical care (UMC) plus chiropractic manipulative therapy
  Medical Care + Chiropractic Care: Patients will receive chiropractic spinal manipulative therapy plus conventional medical care. Medical may include the following: education about self-management, including maintaining activity levels as tolerated and local ice/heat application; pharmacologic management with the use of analgesics and anti-inflammatory agents; and additional therapies that may be applied for volunteers not responding to the initial interventions, including physical therapy and referral to a pain clinic.
- Site: NHP - UMC: Site: Naval Hospital Pensacola
  Conventional medical care only/Usual Medical Care (UMC)
  Conventional Medical Care Only: Conventional medical care may include the following: a focused history and physical examination; limited diagnostic imaging restricted to select volunteers (i.e., for example, those with radiculopathy); education about self-management, including maintaining activity levels as tolerated and local ice/heat application; pharmacologic management with the use of analgesics and anti-inflammatory agents; and additional therapies that may be applied for volunteers not responding to the initial interventions, including physical therapy and referral to a pain clinic.
- Site: NHP - UMC + Chiropractic Care: Site: Naval Hospital Pensacola
  Medical care (UMC) plus chiropractic manipulative therapy
  Medical Care + Chiropractic Care: Patients will receive chiropractic spinal manipulative therapy plus conventional medical care. Medical may include the following: education about self-management, including maintaining activity levels as tolerated and local ice/heat application; pharmacologic management with the use of analgesics and anti-inflammatory agents; and additional therapies that may be applied for volunteers not responding to the initial interventions, including physical therapy and referral to a pain clinic.
- Site: NMCSD - UMC: Site: Naval Medical Center San Diego
  Conventional medical care only/Usual Medical Care (UMC)
  Conventional Medical Care Only: Conventional medical care may include the following: a focused history and physical examination; limited diagnostic imaging restricted to select volunteers (i.e., for example, those with radiculopathy); education about self-management, including maintaining activity levels as tolerated and local ice/heat application; pharmacologic management with the use of analgesics and anti-inflammatory agents; and additional therapies that may be applied for volunteers not responding to the initial interventions, including physical therapy and referral to a pain clinic.
- Site: NMCSD - UMC + Chiropractic Care: Site: Naval Medical Center San Diego
  Medical care (UMC) plus chiropractic manipulative therapy
  Medical Care + Chiropractic Care: Patients will receive chiropractic spinal manipulative therapy plus conventional medical care. Medical may include the following: education about self-management, including maintaining activity levels as tolerated and local ice/heat application; pharmacologic management with the use of analgesics and anti-inflammatory agents; and additional therapies that may be applied for volunteers not responding to the initial interventions, including physical therapy and referral to a pain clinic.
- Total: Total of all reporting groups
Arm/Group | Site: WRNMMC - UMC | Site: WRNMMC - UMC + Chiropractic Care | Site: NHP - UMC | Site: NHP - UMC + Chiropractic Care | Site: NMCSD - UMC | Site: NMCSD - UMC + Chiropractic Care | Total
Number analyzed (Participants) | 125 | 125 | 125 | 125 | 125 | 125 | 750
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (8.4) | 34.7 (8.6) | 25.5 (7.9) | 25.7 (7.5) | 32.4 (7.4) | 32.4 (7.5) | 30.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 19 | 18 | 30 | 29 | 175
  Male | 86 | 85 | 106 | 107 | 95 | 96 | 575
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 9 | 29 | 12 | 21 | 31 | 118
  Not Hispanic or Latino | 109 | 116 | 96 | 113 | 104 | 94 | 632
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 3 | 3 | 1 | 11 | 6 | 30
  Black or African American | 41 | 42 | 17 | 15 | 14 | 20 | 149
  White | 62 | 62 | 102 | 106 | 88 | 87 | 507
  Other or unspecified | 16 | 18 | 2 | 7 | 11 | 17 | 71

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS) for Prior Week
Description: Volunteers will be asked to rate their average level of low back pain (LBP) during the prior week on an ordinal 11-box scale (0=no LBP; 10=worst LBP possible) at baseline and at all of the follow-up assessments. The NRS has excellent metric properties, is easy to administer and score, and has received much use in LBP research. Pain data will be collected at baseline and at all endpoint visits.
Time Frame: Baseline, week 6, week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Site: WRNMMC - UMC | Site: WRNMMC - UMC + Chiropractic Care | Site: NHP - UMC | Site: NHP - UMC + Chiropractic Care | Site: NMCSD - UMC | Site: NMCSD - UMC + Chiropractic Care
Number analyzed (Participants) | 125 | 125 | 125 | 125 | 125 | 125
units on a scale
  Baseline | 4.27 [3.88 to 4.66] | 4.36 [3.98 to 4.75] | 4.73 [4.33 to 5.14] | 4.45 [4.04 to 4.85] | 4.68 [4.28 to 5.08] | 4.87 [4.48 to 5.27]
  Week 6 | 3.90 [3.47 to 4.33] | 3.18 [2.75 to 3.61] | 3.39 [2.92 to 3.85] | 2.17 [1.71 to 2.63] | 4.63 [4.19 to 5.07] | 3.3 [2.86 to 3.74]
  Week 12 | 3.63 [3.18 to 4.07] | 3.21 [2.76 to 3.66] | 2.82 [2.33 to 3.3] | 1.69 [1.2 to 2.17] | 4.0 [3.54 to 4.45] | 2.91 [2.45 to 3.36]
Statistical Analysis 1: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care vs Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care vs Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; All sites combined (week 6) - Between-group differences of mean in LBP; Test type: Superiority; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.4 to -0.7]
Statistical Analysis 2: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care vs Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care vs Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; All sites combined (week 12) - Between-group differences of mean in LBP; Test type: Superiority; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.2 to -0.5]
Statistical Analysis 3: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care; Walter Reed site (week 6) - Between-group differences of mean in LBP; Test type: Superiority; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.3 to -0.1]
Statistical Analysis 4: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care; Walter Reed site (week 12) - Between-group differences of mean in LBP; Test type: Superiority; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.0 to 0.2]
Statistical Analysis 5: Comparison: Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care; Naval Hospital Pensacola site (week 6) - Between-group differences of mean in LBP; Test type: Superiority; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-1.8 to -0.6]
Statistical Analysis 6: Comparison: Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care; Naval Hospital Pensacola site (week 12) - Between-group differences of mean in LBP; Test type: Superiority; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.8 to -0.5]
Statistical Analysis 7: Comparison: Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; Naval Medical Center San Diego site (week 6) - Between-group differences of mean in LBP; Test type: Superiority; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-1.9 to -0.8]
Statistical Analysis 8: Comparison: Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; Naval Medical Center San Diego (week 12) - Between-group differences of mean in LBP; Test type: Superiority; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.7 to -0.5]

2. Primary Outcome: Roland Morris Disability Questionnaire (RMDQ)
Description: We will use a volunteer self-report modified 24-item version of the RMDQ to assess LBP-related disability. The RMDQ may be the most common and respected LBP assessment instrument in LBP outcomes research. It is a one page questionnaire related to LBP disability with documented reliability and validity. It can discriminate between different forms of treatment for back pain, and it is sensitive to clinical change. The RMDQ has been chosen for a number of clinical trials of LBP treatments for its excellent metric properties, ease of use, patient acceptance, and high face validity. This questionnaire will be administered at baseline and at all endpoints. Higher score indicates higher disability. Scale: 0 (no disability) to 24 (maximum disability).
Time Frame: Baseline, week 6, week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Site: WRNMMC - UMC | Site: WRNMMC - UMC + Chiropractic Care | Site: NHP - UMC | Site: NHP - UMC + Chiropractic Care | Site: NMCSD - UMC | Site: NMCSD - UMC + Chiropractic Care
Number analyzed (Participants) | 125 | 125 | 125 | 125 | 125 | 125
units on a scale
  Baseline | 9.94 [8.88 to 11.01] | 9.36 [8.29 to 10.42] | 10.65 [9.52 to 11.78] | 10.21 [9.08 to 11.34] | 8.81 [7.7 to 9.92] | 9.2 [8.08 to 10.32]
  Week 6 | 8.0 [6.8 to 9.19] | 6.22 [5.02 to 7.43] | 5.22 [3.9 to 6.53] | 3.13 [1.83 to 4.43] | 8.8 [7.56 to 10.05] | 6.1 [4.85 to 7.34]
  Week 12 | 7.25 [6.02 to 8.49] | 5.77 [4.52 to 7.02] | 4.4 [3.04 to 5.75] | 2.47 [1.12 to 3.81] | 7.56 [6.29 to 8.84] | 4.83 [3.55 to 6.11]
Statistical Analysis 1: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care vs Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care vs Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; All sites combined (week 6) - RMDQ Between-Group Differences in Disability; Test type: Superiority; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-3.1 to -1.2]
Statistical Analysis 2: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care vs Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care vs Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; All sites combined (week 12) - RMDQ Between-Group Differences in Disability; Test type: Superiority; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-3.0 to -1.0]
Statistical Analysis 3: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care; Walter Reed site (week 6) - RMDQ Between-Group Differences in Disability; Test type: Superiority; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.4 to -0.2]
Statistical Analysis 4: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care; Walter Reed site (week 12) - RMDQ Between-Group Differences in Disability; Test type: Superiority; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-3.2 to 0.2]
Statistical Analysis 5: Comparison: Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care; Pensacola site (week 6) - RMDQ Between-Group Differences in Disability; Test type: Superiority; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-3.8 to -0.4]
Statistical Analysis 6: Comparison: Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care; Pensacola site (week 12) - RMDQ Between-Group Differences in Disability; Test type: Superiority; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-3.7 to -0.2]
Statistical Analysis 7: Comparison: Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; San Diego site (week 6) - RMDQ Between-Group Differences in Disability; Test type: Superiority; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-4.3 to -1.1]
Statistical Analysis 8: Comparison: Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; San Diego site (week 12) - RMDQ Between-Group Differences in Disability; Test type: Superiority; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-4.4 to -1.1]

3. Secondary Outcome: Bothersomeness of Symptoms
Description: The bothersomeness of symptoms commonly associated with LBP will be measured using an existing measure from the LBP literature. Bothersomeness questions are practical and have demonstrated good internal consistency, construct validity, and responsiveness to change with time in patients with LBP and sciatica.
  Possible score ranges from 1 (not at all bothersome) to 5 (extremely bothersome).
Time Frame: Baseline, week 6, week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Site: WRNMMC - UMC | Site: WRNMMC - UMC + Chiropractic Care | Site: NHP - UMC | Site: NHP - UMC + Chiropractic Care | Site: NMCSD - UMC | Site: NMCSD - UMC + Chiropractic Care
Number analyzed (Participants) | 125 | 125 | 125 | 125 | 125 | 125
units on a scale
  Baseline | 3.6 [3.5 to 3.8] | 3.5 [3.3 to 3.6] | 3.7 [3.6 to 3.9] | 3.6 [3.4 to 3.8] | 3.5 [3.3 to 3.6] | 3.4 [3.3 to 3.6]
  Week 6 | 3.0 [2.8 to 3.2] | 2.8 [2.6 to 3.0] | 2.7 [2.4 to 2.9] | 2.1 [1.9 to 2.3] | 3.2 [3.0 to 3.4] | 2.8 [2.6 to 2.9]
  Week 12 | 2.9 [2.7 to 3.1] | 2.8 [2.6 to 3.0] | 2.4 [2.1 to 2.6] | 1.8 [1.6 to 2.1] | 2.9 [2.6 to 3.1] | 2.4 [2.2 to 2.6]
Statistical Analysis 1: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care vs Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care vs Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; All sites combined (week 6) - Between-Group Differences of Means in score of bothersomeness of LBP; Test type: Superiority; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2]
Statistical Analysis 2: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care vs Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care vs Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; All sites combined (week 12) - Between-Group Differences of Means in score of bothersomeness of LBP; Test type: Superiority; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2]
Statistical Analysis 3: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care; Walter Reed site (week 6) - Between-Group Differences of Means in score of bothersomeness of LBP; Test type: Superiority; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 4: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care; Walter Reed site (week 12) - Between-Group Differences of Means in score of bothersomeness of LBP; Test type: Superiority; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1]
Statistical Analysis 5: Comparison: Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care; Pensacola site (week 6) - Between-Group Differences of Means in score of bothersomeness of LBP; Test type: Superiority; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.8 to -0.2]
Statistical Analysis 6: Comparison: Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care; Pensacola site (week 12) - Between-Group Differences of Means in score of bothersomeness of LBP; Test type: Superiority; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.8 to -0.2]
Statistical Analysis 7: Comparison: Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; San Diego site (week 6) - Between-Group Differences of Means in score of bothersomeness of LBP; Test type: Superiority; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.7 to -0.2]
Statistical Analysis 8: Comparison: Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; San Diego site (week 12) - Between-Group Differences of Means in score of bothersomeness of LBP; Test type: Superiority; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.7 to -0.1]

4. Secondary Outcome: Numerical Pain Rating Scale (NRS) for Past 24 Hours
Description: Volunteers will be asked to rate their level of pain on that day on an ordinal 11-box scale (0=no LBP; 10=worst LBP possible) at baseline and at all of the follow-up assessments. The NRS has excellent metric properties, is easy to administer and score, and has received much use in LBP research. Pain data will be collected at baseline and at all endpoint visits. The question will capture information pertaining to pain over the last 24 hours.
Time Frame: Baseline, week 6, week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Site: WRNMMC - UMC | Site: WRNMMC - UMC + Chiropractic Care | Site: NHP - UMC | Site: NHP - UMC + Chiropractic Care | Site: NMCSD - UMC | Site: NMCSD - UMC + Chiropractic Care
Number analyzed (Participants) | 125 | 125 | 125 | 125 | 125 | 125
units on a scale
  Baseline | 5.4 [5.2 to 5.7] | 5.6 [5.4 to 5.8] | 6.1 [5.9 to 6.4] | 5.9 [5.6 to 6.1] | 5.4 [5.2 to 5.6] | 5.4 [5.2 to 5.6]
  Week 6 | 4.5 [4.1 to 5.0] | 3.9 [3.4 to 4.3] | 3.4 [2.9 to 3.9] | 2.1 [1.6 to 2.6] | 5.3 [4.8 to 5.7] | 3.6 [3.2 to 4.1]
  Week 12 | 4.4 [3.9 to 4.9] | 3.7 [3.2 to 4.2] | 3.0 [2.4 to 3.5] | 1.4 [0.9 to 2.0] | 4.3 [3.8 to 4.8] | 3.2 [2.7 to 3.7]
Statistical Analysis 1: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care vs Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care vs Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; All sites combined (week 6) - NRS score for worst LBP in past 24 hours - Between-Group Differences of Mean; Test type: Superiority; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-1.6 to -0.8]
Statistical Analysis 2: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care vs Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care vs Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; All sites combined (week 12) - NRS score for worst LBP in past 24 hours - Between-Group Differences of Mean; Test type: Superiority; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.6 to -0.7]
Statistical Analysis 3: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care; Walter Reed site (week 6) - NRS score for worst LBP in past 24 hours - Between-Group Differences of Mean; Test type: Superiority; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.3 to -0.02]
Statistical Analysis 4: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care; Walter Reed site (week 12) - NRS score for worst LBP in past 24 hours - Between-Group Differences of Mean; Test type: Superiority; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.5 to -0.1]
Statistical Analysis 5: Comparison: Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care; Pensacola site (week 6) - NRS score for worst LBP in past 24 hours - Between-Group Differences of Mean; Test type: Superiority; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.0 to -0.7]
Statistical Analysis 6: Comparison: Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care; Pensacola site (week 12) - NRS score for worst LBP in past 24 hours - Between-Group Differences of Mean; Test type: Superiority; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-2.3 to -0.8]
Statistical Analysis 7: Comparison: Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; San Diego site (week 6) - NRS score for worst LBP in past 24 hours - Between-Group Differences of Mean; Test type: Superiority; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-2.3 to -1.0]
Statistical Analysis 8: Comparison: Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; San Diego site (week 12) - NRS score for worst LBP in past 24 hours - Between-Group Differences of Mean; Test type: Superiority; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-1.9 to -0.5]

5. Secondary Outcome: Healthcare Utilization & Medication Use
Description: Based on the pilot study, volunteers will most likely have been seen by other healthcare providers and prescribed pain medication by a primary care provider prior to being enrolled in the study, this questionnaire will ensure that we collect all healthcare and medication use.
Time Frame: week 6, week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Site: WRNMMC - UMC | Site: WRNMMC - UMC + Chiropractic Care | Site: NHP - UMC | Site: NHP - UMC + Chiropractic Care | Site: NMCSD - UMC | Site: NMCSD - UMC + Chiropractic Care
Number analyzed (Participants) | 125 | 125 | 125 | 125 | 125 | 125
Participants
  Week 6 Med Frequency: 0 days | 25 | 36 | 28 | 34 | 39 | 40
  Week 6 Med Frequency: 1-2 days | 20 | 24 | 12 | 17 | 22 | 20
  Week 6 Med Frequency: 3-4 days | 13 | 7 | 10 | 1 | 12 | 8
  Week 6 Med Frequency: 5-6 days | 8 | 8 | 1 | 3 | 10 | 9
  Week 6 Med Frequency: 7 days | 14 | 8 | 11 | 8 | 9 | 8
  Week 6 Med Frequency: missing | 45 | 42 | 63 | 62 | 33 | 40
  Week 12 Med Frequency: 0 days | 26 | 38 | 38 | 48 | 49 | 42
  Week 12 Med Frequency: 1-2 days | 23 | 15 | 7 | 5 | 21 | 23
  Week 12 Med Frequency: 3-4 days | 9 | 12 | 7 | 4 | 10 | 7
  Week 12 Med Frequency: 5-6 days | 10 | 1 | 4 | 2 | 4 | 5
  Week 12 Med Frequency: 7 days | 12 | 17 | 6 | 4 | 8 | 8
  Week 12 Med Frequency: missing | 45 | 42 | 63 | 62 | 33 | 40
Statistical Analysis 1: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care vs Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care vs Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; Week 6: All 3 sites combined; Test type: Superiority; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.54 to 0.97]
Statistical Analysis 2: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care vs Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care vs Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; Week 12: All 3 sites combined; Test type: Superiority; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.58 to 1.0]

6. Secondary Outcome: Global Improvement Scale
Description: This is a modification of the visual analog scale (VAS) developed to assess degree of improvement over a specified period of time. Global low back pain (LBP) improvement was assessed by asking participants to rate their perceived LBP improvement since baseline on a 7-point scale: 0 = completely gone, 1 = much better, 2 = moderately better, 3 = a little better, 4 = about the same, 5 = a little worse, 6 = much worse.
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Groups:
- WR - UMC: Walter Reed National Military Medical Center (WR) - Usual Medical Care
- WR - UMC + CC: Walter Reed National Military Medical Center - Usual Medical Care + Chiropractic Care group
- Pensacola - UMC: Naval Hospital Pensacola - Usual Medical Care group
- Pensacola - UMC + CC: Naval Hospital Pensacola - Usual Medical Care + Chiropractic Care group
- San Diego - UMC: Naval Medical Center San Diego - Usual Medical Care group
- San Diego - UMC + CC: Naval Medical Center San Diego - Usual Medical Care + Chiropractic Care group
Arm/Group | WR - UMC | WR - UMC + CC | Pensacola - UMC | Pensacola - UMC + CC | San Diego - UMC | San Diego - UMC + CC
Number analyzed (Participants) | 125 | 125 | 125 | 125 | 125 | 125
Participants
  Completely gone | 1 | 2 | 7 | 16 | 0 | 4
  Much better | 12 | 26 | 20 | 32 | 10 | 22
  Moderately better | 9 | 23 | 9 | 11 | 4 | 15
  A little better | 12 | 20 | 11 | 7 | 8 | 22
  About the same | 37 | 18 | 15 | 5 | 47 | 26
  A little worse | 15 | 2 | 8 | 1 | 23 | 5
  Much worse | 3 | 2 | 1 | 1 | 6 | 0
  missing | 36 | 32 | 54 | 52 | 27 | 31
Statistical Analysis 1: Comparison: WR - UMC vs WR - UMC + CC vs Pensacola - UMC vs Pensacola - UMC + CC vs San Diego - UMC vs San Diego - UMC + CC; All sites combined: 6 weeks; Test type: Superiority; Odds Ratio (OR) = 0.18, 95% CI 2-sided [0.13 to 0.25]
Statistical Analysis 2: Comparison: WR - UMC vs WR - UMC + CC; Walter Reed site: 6 weeks; Test type: Superiority; Odds Ratio (OR) = 0.26, 95% CI 2-sided [0.16 to 0.42]
Statistical Analysis 3: Comparison: Pensacola - UMC vs Pensacola - UMC + CC; Naval Hospital Pensacola site: 6 weeks; Test type: Superiority; Odds Ratio (OR) = 0.18, 95% CI 2-sided [0.10 to 0.33]
Statistical Analysis 4: Comparison: San Diego - UMC vs San Diego - UMC + CC; Naval Medical Center San Diego site: 6 weeks; Test type: Superiority; Odds Ratio (OR) = 0.13, 95% CI 2-sided [0.08 to 0.21]

7. Secondary Outcome: Patient Satisfaction
Description: A one item patient satisfaction questionnaire. Satisfaction is measured as means on a numerical rating scale, 0 [not at all satisfied] to 10 [extremely satisfied].
Time Frame: Week 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Site: WRNMMC - UMC | Site: WRNMMC - UMC + Chiropractic Care | Site: NHP - UMC | Site: NHP - UMC + Chiropractic Care | Site: NMCSD - UMC | Site: NMCSD - UMC + Chiropractic Care
Number analyzed (Participants) | 125 | 125 | 125 | 125 | 125 | 125
units on a scale | 5.65 [5.19 to 6.11] | 7.64 [7.17 to 8.11] | 6.04 [5.51 to 6.56] | 8.34 [7.82 to 8.85] | 4.34 [3.86 to 4.83] | 7.45 [6.97 to 7.93]
Statistical Analysis 1: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care vs Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care vs Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; All sites combined: 6 weeks; Test type: Superiority; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [2.1 to 2.8]
Statistical Analysis 2: Comparison: Site: WRNMMC - UMC vs Site: WRNMMC - UMC + Chiropractic Care; Walter Reed site: 6 weeks; Test type: Superiority; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [1.4 to 2.6]
Statistical Analysis 3: Comparison: Site: NHP - UMC vs Site: NHP - UMC + Chiropractic Care; Naval Hospital Pensacola site: 6 weeks; Test type: Superiority; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [1.6 to 3.0]
Statistical Analysis 4: Comparison: Site: NMCSD - UMC vs Site: NMCSD - UMC + Chiropractic Care; Naval Medical Center San Diego site: 6 weeks; Test type: Superiority; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [2.5 to 3.7]

8. Secondary Outcome: Patient Expectation
Description: Previous work has shown that patient expectation regarding benefit of care can be a significant non-specific effect.
  The score indicates participant's expectation of helpfulness of treatment for LBP, measured on a scale of 0 (not helpful at all) to 10 (extremely helpful).
Time Frame: Baseline only
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Sites - UMC: All 3 sites combined (WRNMMC, NHP, NMCSD)
  Conventional medical care only/Usual Medical Care (UMC)
  Conventional Medical Care Only: Conventional medical care may include the following: a focused history and physical examination; limited diagnostic imaging restricted to select volunteers (i.e., for example, those with radiculopathy); education about self-management, including maintaining activity levels as tolerated and local ice/heat application; pharmacologic management with the use of analgesics and anti-inflammatory agents; and additional therapies that may be applied for volunteers not responding to the initial interventions, including physical therapy and referral to a pain clinic.
- All Sites Combined - UMC + Chiropractic Care: All 3 sites combined (WRNMMC, NHP, NMCSD)
  Medical care (UMC) plus chiropractic manipulative therapy
  Medical Care + Chiropractic Care: Patients will receive chiropractic spinal manipulative therapy plus conventional medical care. Medical may include the following: education about self-management, including maintaining activity levels as tolerated and local ice/heat application; pharmacologic management with the use of analgesics and anti-inflammatory agents; and additional therapies that may be applied for volunteers not responding to the initial interventions, including physical therapy and referral to a pain clinic.
Arm/Group | Site: WRNMMC - UMC | Site: WRNMMC - UMC + Chiropractic Care | Site: NHP - UMC | Site: NHP - UMC + Chiropractic Care | Site: NMCSD - UMC | Site: NMCSD - UMC + Chiropractic Care | All Sites - UMC | All Sites Combined - UMC + Chiropractic Care
Number analyzed (Participants) | 125 | 125 | 125 | 125 | 125 | 125 | 750 | 750
units on a scale
  Expectation UMC + Chiropractic Care | 8.2 (1.8) | 8.4 (1.6) | 8.1 (1.9) | 8.3 (1.9) | 8.6 (1.8) | 8.5 (1.9) | 8.3 (1.9) | 8.4 (1.8)
  Expectation UMC | 5.3 (2.4) | 4.9 (2.5) | 5.3 (2.3) | 5.4 (2.5) | 4.5 (2.8) | 5.2 (3.0) | 5.0 (2.5) | 5.2 (2.7)

9. Secondary Outcome: Back Pain Functional Scale (BPFS)
Description: The BPFS is a 12-question functional status survey designed for use as an individual patient decision-making tool. Each of the 12 questions is answered using a 5-point Likert-type scale and therefore scores for this scale will range from 0-60 (higher scores indicate better function). In recent studies, the BPFS is improved sensitivity to change than the RMDQ. This scale will be administered at baseline and all endpoint visits.
Time Frame: Baseline and all endpoint visits (week 2, week 4, week 6, week 12)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Site: WRNMMC - UMC | Site: WRNMMC - UMC + Chiropractic Care | Site: NHP - UMC | Site: NHP - UMC + Chiropractic Care | Site: NMCSD - UMC | Site: NMCSD - UMC + Chiropractic Care
Number analyzed (Participants) | 125 | 125 | 125 | 125 | 125 | 125
units on a scale
  Baseline | 39.48 [37.5 to 41.47] | 39.18 [37.2 to 41.16] | 37.68 [35.57 to 39.78] | 38 [35.9 to 40.1] | 39.97 [37.9 to 42.03] | 39.98 [37.9 to 42.06]
  Week 2 | 42.08 [39.92 to 44.23] | 42.65 [40.52 to 44.7] | 44.21 [41.81 to 46.59] | 46.76 [44.46 to 49.06] | 39.07 [36.87 to 41.28] | 42.45 [40.24 to 44.66]
  Week 4 | 42.03 [39.76 to 44.3] | 44.77 [42.49 to 47.04] | 46.45 [43.93 to 48.97] | 50.31 [47.87 to 52.76] | 39.36 [37.03 to 41.68] | 45.02 [42.69 to 47.35]
  Week 6 | 42.72 [40.47 to 44.96] | 45.74 [43.5 to 47.98] | 48.55 [46.06 to 51.04] | 52.64 [50.21 to 55.08] | 40.52 [38.2 to 42.83] | 46.02 [43.72 to 48.32]
  Week 12 | 43.73 [41.43 to 46.03] | 45.51 [43.2 to 47.82] | 49.7 [47.15 to 52.25] | 54.56 [52.04 to 57.07] | 43.57 [41.23 to 45.91] | 47.8 [45.46 to 50.15]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Any untoward medical occurence that may present itself during the conduct of the study which may or may not have a causal relationship with the study procedures.
  *The total number of Adverse Events (AEs) may exceed the total # of people affected because some people experienced multiple AEs.
  AEs were monitored via self-report AE collected at Week 2, Week 4, and Week 6 assessments or via self-report to the study physician or site project manager directly during the 12 week period.
Groups:
- Usual Medical Care: Conventional medical care only/usual medical care (UMC)
  Conventional Medical Care Only: Conventional medical care may include the following: a focused history and physical examination; limited diagnostic imaging restricted to select volunteers (i.e., for example, those with radiculopathy); education about self-management, including maintaining activity levels as tolerated and local ice/heat application; pharmacologic management with the use of analgesics and anti-inflammatory agents; and additional therapies that may be applied for volunteers not responding to the initial interventions, including physical therapy and referral to a pain clinic.
- UMC + Chiropractic Care: Medical care plus chiropractic manipulative therapy
  Medical Care + Chiropractic Care: Patients will receive chiropractic spinal manipulative therapy plus conventional medical care. Medical may include the following: education about self-management, including maintaining activity levels as tolerated and local ice/heat application; pharmacologic management with the use of analgesics and anti-inflammatory agents; and additional therapies that may be applied for volunteers not responding to the initial interventions, including physical therapy and referral to a pain clinic.
Arm/Group | Usual Medical Care | UMC + Chiropractic Care
All-Cause Mortality (participants affected / at risk) | 0/375 | 0/375
Serious Adverse Events (participants affected / at risk) | 0/375 | 0/375
Other Adverse Events (participants affected / at risk) | 13/375 | 33/375
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Medical Care (N=375) | UMC + Chiropractic Care (N=375)
Spine-related pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 24 (30)
Spine-related pain with radiation (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (5)
Extremity pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
General stiffness/tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscle spasm/cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No